CLINICAL TRIAL: NCT01156740
Title: Treatment of Pharyngitis Study (TOPS): A Randomized Equivalence Trial of Intramuscular Penicillin G vs. Oral Amoxicillin Antibiotics for the Treatment of Streptococcal Pharyngitis in Children in Developing Countries
Brief Title: Treatment of Group A Beta Hemolytic Streptococcal Pharyngitis in Children in Low Resource Settings
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); World Health Organization (Other); Cairo University (Other); University Hospital for Infectious Diseases, Croatia (Other); Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Dr. Mark C. Steinhoff, Cincinnati Children's Hospital / Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRN-A-00-96-90006-00
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2009-12

CONDITIONS: Streptococcal Infections; Pharyngitis
Keywords: streptococcal pharyngitis; randomized clinical trial; amoxicillin; intramuscular benzathine penicillin G.
MeSH Terms: conditions — Streptococcal Infections; Pharyngitis | interventions — Penicillin G; beta Lactam Antibiotics; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intramuscular benzathine Penicillin G (Active Comparator): A single dose of intramuscularly administered intramuscular benzathine penicillin G (IM BPG). The dosing was as follows: IM BPG; 600,000 U > 27kg or 1,200,000 U <27 kg
  Interventions: Drug: Penicillin G, Benzathine
- Amoxicillin (Active Comparator): A 10-day once daily dose of Amoxicillin was given in an oral form. The first dose was given at the time of randomization, and parents were instructed on giving the remaining doses. Dosing was as follows: 750 mg/QD
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Penicillin G, Benzathine — IM BPG; 600,000 U > 27kg or 1,200,000 U <27 kg)
  Other Names: Intramuscular Benzathine Penicillin G; Beta-lactam antibiotics
  Arms: Intramuscular benzathine Penicillin G
Drug: Amoxicillin — 750 mg/QD
  Other Names: Amoxil®; Trimox®
  Arms: Amoxicillin

SUMMARY:
The purpose of this study was to compare the microbiological effects of two different treatments: a single dose of intramuscular benzathine penicillin G (IM BPG) vs. a 10-day daily dose of amoxicillin for the treatment of GABHS pharyngitis in children in low resource settings. This study was a prospective multi-center randomized active control treatment trial. The trial is a non-inferiority equivalence trial, to determine if amoxicillin treatment is at least as effective as the currently given IM BPG treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-12 years old,
* Presenting with complaint of sore throat
* Parental consent given and child assent if 5 years or older

Exclusion Criteria:

* The parent/guardian reported oral antibiotic use in the past 3 days or injectable penicillin in past 28 days prior to screening
* Had a history of rheumatic fever or rheumatic heart disease
* Required hospitalization for any reason at the time of enrollment
* Had previously been enrolled in the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 558 (Actual)
Dates: Start 2001-08; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Eradication of Group A Streptococcus (GAS) | 21-28 days after 1st visit
  The primary outcome of the study was bacteriologic treatment success, which was defined as eradication of GAS from the pharynx at the follow up visit. Eradication was defined as no GAS present on the throat culture.

SECONDARY OUTCOMES:
Compliance to treatment | 21-28 days after 1st visit
  Compliance with the amoxicillin treatment regimen was assessed at the follow up visit. The primary measure of compliance was the presence of antimicrobial activity in the urine-impregnated filter paper strips. For those who did not return the filter paper strip, compliance was measured by parent/guardian report during the exit interview. Patients who did not fulfill at least one of these criteria were considered noncompliant.

CONTACTS AND LOCATIONS:
Overall Officials: Mark C. Steinhoff, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Federal University of Rio de Janeiro, Rio de Janeiro, Brazil
- University Hospital for Infectious Diseases, Zagreb, Croatia
- Cairo University, Cairo, Egypt